CLINICAL TRIAL: NCT05412615
Title: Proximal Row Carpectomy With Meniscal Allograft Arthroplasty for Wrist Osteoarthritis
Brief Title: PRC With Meniscal Allograft Arthroplasty for Wrist Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 21-3148
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Wrist Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meniscal Allograft with PRC (Experimental): These patients will receive a tissue allograft with their wrist reconstruction procedure.
  Interventions: Procedure: Meniscus Allograft Transplantation with Proximal Row Carpectomy
- PRC only (Placebo Comparator): These patients will receive the standard proximal row carpectomy procedure.
  Interventions: Procedure: Proximal Row Carpectomy

INTERVENTIONS:
Procedure: Meniscus Allograft Transplantation with Proximal Row Carpectomy — Supplementing the wrist reconstruction with a meniscal allograft to improve wrist function and pain scores.
  Arms: Meniscal Allograft with PRC
Procedure: Proximal Row Carpectomy — Standard proximal row carpectomy with no tissue or synthetic adjuncts
  Arms: PRC only

SUMMARY:
This study plans to learn more about the effect of adding tissue graft for wrist osteoarthritis reconstruction procedures. Previous studies have shown better allograft stability, and no documented foreign body reaction than with silicone and other synthetic materials.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic wrist arthritis associated with SLAC or SNAC pathology
* Patients 30 years or older or 80 years or younger

Exclusion Criteria:

* Patients younger than 29 years or older than 80 years
* History of previous surgery related to wrist osteoarthritis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: Baseline/Pre-op | Preoperatively
  Participant wrist disability score will be assessed before and after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 2 weeks | 2 weeks
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 6 weeks | 6 weeks
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 3 months | 3 months
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 6 months | 6 months
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 9 months | 9 months
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 12 months | 12 months
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.
DISABILITIES OF THE ARM, SHOULDER AND HAND Score: 24 months | 24 months
  Participant wrist disability score after their wrist reconstruction procedure. Disability of the arm, shoulder and hand (DASH) score ranges from (0-100) with higher score being worse and representing more disability. Lower scores are better and represent less disability. The questionnaire contains 11 questions about daily tasks which are rated 1 (no difficulty) to 5 (Unable to perform) for each question.

SECONDARY OUTCOMES:
Pain Score | Preoperatively, up to 24 Months
  Visual Analog Pain Score
Radiographic joint spacing | 3 months, up to 24 Months
  Measurement of joint spacing in the wrist in millimeters.
MRI Joint Spacing | 9 Months, 24 Months
  Wrist joint spacing measurements in millimeters using Magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- UCHealth Steadman Hawkins Clinic Inverness, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No